# **Protocol Document**

ClinicalTrials.gov Identifier: NCT05187013

Unique Protocol ID: NCR203140

Title: mHealth to Address Uncontrolled Hypertension Among Hypertensive Homeless Adults

Version Date: January 26, 2021

### STUDY PROTOCOL

## **Project Summary**

Annually, millions of Americans experience homelessness. Hypertension (HTN) is one of the most common conditions among persons experiencing homelessness (PEH) but is often uncontrolled; 40.1% of hypertensive PEH have uncontrolled blood pressure (BP) compared to 24.8% of hypertensive adults in the general population. PEH face multiple barriers to therapeutic lifestyle changes that complicate their HTN management. Strategies targeting self-management behaviors and counseling to support adherence to medications and lifestyle changes contribute to better BP control and significant cardiovascular risk reduction. However, these strategies are not available or accessible to the PEH. At the patient level, educational interventions with behavioral support through continued patient contact over months are effective in the treatment of chronic diseases including HTN. The mHealth strategies including short messaging service (SMS) texting have been shown to improve adherence to BP medications and BP control and were feasible and acceptable among hypertensive adults. Majority of the PEH have access to mobile phones that can receive and send SMS texts. Considering mobility of the PEH, we propose that an mHealth strategy using SMS texting could be used as a platform for better communication and information management for BP control, facilitate coordination of care, support behavior changes, and improve targeted outreach. The mHealth strategies for HTN have never been evaluated in the PEH despite the growing evidence of their effectiveness and the accessibility of mobile phones among PEH. This study will test this strategy and pave the way for its utilizations in the health settings where the PEH seek care and has potentials for adaptation for control of other chronic diseases among PEH. This study will be implemented in shelter-clinics in New York City (NYC) and in collaboration with community organizations making sustainability of the intervention effects and its scalability feasible. We propose a mixed methods study: AIM1: To evaluate the efficacy of a 6-month SMS texting targeted on HTN management (INT) versus an attention control (CL) on changes in systolic BP (SBP) and diastolic BP (DBP) and adherence to BP medications and appointments at 6 months in hypertensive PEH with uncontrolled BP age 21 or older (n=120). H1) Those randomized to the INT (n=60) will exhibit at least 8 mmHg reduction in either SBP or DBP compared to those randomized to the CL (n=60) at 6 months. H2) The INT group will exhibit better adherence to BP medications and appointments compared to those in the CL at 6 months. BP readings and adherence to appointments and medications will be measured at regular clinic visits. Randomization will be at the individual level in the shelter-clinics. AIM2: To assess patients' and providers' attitudes, acceptability, and experience of a 6-month mHealth SMS texting for HTN management in hypertensive PEH age 21 or older with uncontrolled BP in NYC's shelter-clinics. We will use semi-structured interviews using random and criteria sampling of the PEH and providers.

### **APPROACH**

Overview of study design and intervention: Participants will be recruited directly in the clinics, via medical record reviews, and through the outreach team. Individual participants will be assigned to treatment groups by a computer-assisted permuted randomization schedule using of a block size of four, stratified by clinic site (n=2) a. Inclusion criteria: patient PEH age 21 or older already diagnosed with HTN whose SBP or DBP at the most recent clinic visit were >140 or >90 mmHg, respectively (see Clinic Visits) (54); English or Spanish speaking; currently presenting to the PR shelter-clinics for medical care; connected to multidisciplinary social and health services in the PR. Exclusion criteria: pregnant or within three months postpartum (55); recent heart attack or stroke (in the previous 6 months); aortic aneurysm, end stage renal disease or on dialysis; inability to read and respond to SMS texts; severe mental illness; current severe or uncontrolled substance abuse or any condition preventing participants to provide informed consent. Patients with a SBP >175 mmHg or DBP >105 are eligible only if they have no symptoms suggesting a hypertensive emergency or urgency evaluated by a medical provider (55). In these cases, providers will be given notification of intent to enroll the patient in this study and have 48 hours to opt them out of the study for any reason including mental and physical health issues. Provider participants are PR's physicians, NPs, social workers, counselors working at the sites not involved in study design or implementation. The intervention will include 6 months of mHealth HTN management support via SMS texts including reminders for medication adherence, appointment attendance, and HTN specific health education and support. The control group will receive 6

months of mHealth including basic healthcare and general health promotion via SMS texts. Both groups undergo BP measurements and adherence assessment at regular clinic visits. Participants will have a follow-up appointment scheduled at 2 months by the research associate at the baseline visit. Data obtained from patients via SMS texts is reviewed by the system and study team members. During the study, feedback to SMS texts, including automated and reciprocal feedback responding to patient-specific input, will be directly provided to the patients within the same day to enhance education and behavioral changes in a protocolized fashion. We will recruit a total of PEH (n=120) with uncontrolled HTN and a range of providers from the PR in NYC. The timeline will consist of socio-demographics and baseline data collected at the enrollment followed by a 6-month mHealth for each participant until the last enrolled participant completes the study. Primary outcomes of BP readings, medication adherence (Voils DOSE-nonadherence (68,69)), and appointment attendance will be measured at regular clinic visits. Other outcomes include phone retention rates; utilization of phones and SMS texts (# of texts read and responded by subjects). PEH with HTN and providers will be interviewed. Research assistants (RA), fluent in Spanish, will perform semi-structured interviews and collect data. Interim analysis will be performed; the final analysis of quantitative and qualitative data will ensue after the completion of data collection.

Study Procedures: Hypertensive PEH with uncontrolled BP will be identified and enrolled from the proposed site during weekdays via both electronic medical records and during their clinic visit on the day of enrollment and will be approached in the waiting rooms and offered to participate in the study. Potential unsheltered participants' eligibility will be assessed at the two predetermined clinic sites.. Uncontrolled BP is measured by the BP readings from the most recent visit (Clinic Visit below) and defined based on the current updated guideline and diagnoses of HTN. (54) Patient's other co-morbidities (CAD, stroke, MI, DM or chronic kidney disease) will be collected but will not be factored into eligibility assessment. The study is described to potential participants as "a study to evaluate the effect of mobile technology/SMS texts on improving HTN control for persons experiencing homelessness". If accepted, participants will be consented in a private area/room. Participants with severe mental illness or current severe or uncontrolled substance abuse will be excluded. Socio-demographics and baseline data will be collected including BP measurements by clinic nurses, and behavioral surveys, medication adherence measurements, and other data by RA. RA will offer health education on HTN for 20 minutes to all participants; provide them with free single type of cell phones (with calendar and WiFi access) with unlimited minutes and text plans for the study period; train them how to charge and maintain phones and use SMS texts; and provide ongoing help and follow-ups to assure proper understanding and usage of the phones. Lost/broken phones are replaced free of charge. At enrollment, participants will be randomly assigned to either the INT or CL group described above. Study coordinator will oversee randomization and supervise the application and implementation of the mHealth.

Brief description of mHealth/SMS texting, technology requirement, and communication venues: In initial phase of this study, to better develop and adapt the intervention, we will use a community-based participatory approach to incorporate views from a group of hypertensive PEH, shelter case workers, counselors, and providers. Using focus groups, we will explore literacy factors, HTN health literacy, and mobile technology literacy to adapt SMS platform, the intervention and its components, and evaluation tools. This process will also help further understand and address chronic diseases among other priorities. The study's AIM 1 will also help understand challenges and opportunities and refine the intervention for subsequent studies. In the INT group, participants will receive SMS texts every other day (58) to reinforce medication and appointment adherence, lifestyle changes, and health promotions related to HTN control and CVD risks. For appointment adherence, they will receive reminder SMS texts, 3 and 1 days before each appointment, with a follow up text if missed the appointment. SMS text queries will also be sent about PB medications' side effects. Texts are interactive and reciprocal; for example, if patients send texts (helping in refill medications, answering specific medication, nutrition or other questions) they will be responded within the same day by the system, or directed to an NP and or referred to the PI if need further help. For urgent matters, RA and study coordinator will direct patients to clinic providers or emergency room. If there is no response from participants after one week/three texts, the study coordinator will call to help troubleshoot or address potential reasons for dropouts. We have already identified technology companies to provide the SMS platform (English & Spanish) and IT development services for this study; evaluated their HTN management SMS platforms; and will further adapt and modify them for the intervention and attention control arms. Participants in both groups will receive welcome texts

(Thank you for participating. We will never ask for personal/banking details. Participation is voluntary etc.) and Birthday SMS-texts. Tables 1 presents brief constructs and examples of SMS texts in the INT group (29,55,59).

Table 1. Examples of intervention group's SMS texts for medication adherence in English for each construct (29,55,59)

| Self-efficacy | "Have you taken all your medications in the past? Write down what helped you be successful" |
|---|---|
| Motivation | "Set a short-term goal, and achieve it! "You will do whatever it takes to take your medications as prescribed" |
| Social Support | "Ask someone you trust to help you remember to take your medicine as directed" |
| Importance | "Blood pressure can't be cured. To keep healthy, keep on with your pills" "What would you say to your loved ones if they were not taking their medications? Say it to yourself" |
| Knowledge, attitude, barriers | "Use a pillbox to organize your medications" "Talking to your doctor or pharmacist about your medications helps you understand why you are taking them" "Leave yourself a note, voice or email to take medications" |
| Implementation,<br>Intention | "Make taking your pills part of your daily routine, like brushing teeth. It helps take them regularly" "If I have 5 pills left in my bottle, I will call the pharmacy for a refill" "Going on a trip, I will pack my medicine first!" |

The CL arm will receive SMS texts regarding basic general health and health promotions such as the importance of hydration (58), and safety and protection that do not overlap with HTN specific management. The INT arm also receives the same basic general health texts. Both groups will receive routine robocalls regarding their appointments and if they missed them. IT company services will be free of charge for subjects. Clinic Visits: After enrollment, participants will be scheduled for assessment visits in the shelter-clinics to measure and record their BP readings and medication adherence at regular clinic visits. They will continue to have regular care with their respective providers at their clinics. Blood pressure is measured by clinic nurses at the initial enrollment and at each follow-ups to the end of study follow-up period for each participant. Measurements will be taken per clinic protocols for proper blood pressure measurements (60). Since patients are already diagnosed with HTN, BP readings from the most recent visit will be used to determine uncontrolled vs controlled HTN. Uncontrolled BP is defined based on the current updated guideline (SBP>140 or DPB>90 mmHq) (54). If BP readings indicate critical values, a clinic medical provider will evaluate the patient as an urgent visit and offer the appropriate care. For medication adherence, at each assessment visits, Volis DOSenonadherence will be used. Since this population has unstable housing, unannounced pill counts are not feasible. Appointment attendance will be measured by accessing medical records. At enrollment, we will collect socio-demographics and clinical data including age, race/ethnicity, gender, years and episodes of homelessness, BMI, health insurance status, and history of chronic disease (diabetes, renal insufficiency, hyperlipidemia, asthma, COPD and CAD/MI, tobacco, alcohol or substance abuse, or mental illness). Attrition/Retention: Clients at PR on average stay 1 year within the system which will decrease the attrition rate as they will be reachable in shelters; many patients continue to see their providers afterward. If no responses to texts in one week/three texts, the study coordinator will contact patients by phone and seek support from shelters case workers to connect and identify and address issues related to drop out. Multidisciplinary teams in the shelters to address social barriers and improve social services will help decrease drop-outs.

**Data Management**: All data received via SMS texting will be captured through the SMS texting interface developed for this project. Each enrolled participant will have a unique identifying ID that will capture their baseline and ongoing outcome data as entered by the RA. All data will be collected and sent electronically in password-encrypted files via an electronic cloud-based system to the GWU data management team that maintain and managed them. The data will be reviewed on a bimonthly basis and issues will be communicated to the contact PI to be addressed during the coordinator's periodic visits to the sites. Outlying, inconsistent data, and missing data will be the targets of the data quality review.

**Timeline:** Coordination of research & IRB (Mon 1-3); mHealth development and implementation (Mon 1-5); Recruitment and ongoing enrollment, data collection and patient interviews (Mon 6-18); Providers' qualitative interviews (Mon 18-20); Data cleaning and analyses, manuscripts preparation for dissemination (Mon 7-24).

### Reference:

- 1. National Alliance to End Homelessness. The State of Homelessness in America 2020. (accessed June 2, 2020). Available at https://endhomelessness.org/homelessness-in-america/homelessness-statistics/state-ofhomelessness-2020
- 2. National Alliance to End Homelessness. The State of Homelessness in America 2013. Homeless Research Institute. Accessed June 2 2020, available at http://www.ncdsv.org/images/NAEH StateOfHomelessnessInAmerica 4-2013.pdf
- 3. Fargo J, Metraux S, Byrne T, Munley E, Montgomery AE, Jones H, Sheldon G, Kane V, Culhane D. Prevalence and Risk of Homelessness Among US Veterans. Prev Chronic Dis. 2012; 9: E45. Epub 2012 Jan 26.
- 4. Culhane DP, Metraux S, Byrne T, Stino M, Bainbridge J. The age structure of contemporary homelessness: evidence and implications for public policy. Analyses of Social Issues and Public Policy, 2013 Jan, DOI:10.1111/asap.12004. available at <a href="https://spssi.onlinelibrary.wiley.com/doi/abs/10.1111/asap.12004">https://spssi.onlinelibrary.wiley.com/doi/abs/10.1111/asap.12004</a>
- 5. Kushel MB, Vittinghoff E, Haas JS. "Factors associated with the health care utilization of homeless persons." JAMA. 2001 Jan 10;285(2):200-6.
- 6. Bernstein, R. S., Meurer, L. N., Plumb, E. J., & Jackson, J. L. Diabetes and hypertension prevalence in homeless adults in the United States: a systematic review and meta-analysis. Am J Public Health, 2015;105(2): e46-e60.
- 7. Gelberg L1, Linn LS. Assessing the physical health of homeless adults. JAMA. 1989 Oct 13;262(14):1973-9.
- 8. Szerlip MI1, Szerlip HM. dentification of cardiovascular risk factors in homeless adults. Am J Med Sci. 2002 Nov;324(5):243-6.
- 9. Moczygemba LR1, Kennedy AK, Marks SA, Goode JV, Matzke GR. A qualitative analysis of perceptions and barriers to therapeutic lifestyle changes among homeless hypertensive patients. Res Social Adm Pharm. 2013 Jul-Aug;9(4):467-81. doi: 10.1016/j.sapharm.2012.05.007. Epub 2012 Jul 25.
- Kim DH1, Daskalakis C, Plumb JD, Adams S, Brawer R, Orr N, Hawthorne K, Toto EC, Whellan DJ. Modifiable cardiovascular risk factors among individuals in low socioeconomic communities and homeless shelters. Fam Community Health. 2008 Oct-Dec;31(4):269-80. doi: 10.1097/01.FCH.0000336090.37280.2e.
- 11. Savage CL1, Lindsell CJ, Gillespie GL, Dempsey A, Lee RJ, Corbin A. Health care needs of homeless adults at a nurse-managed clinic. J Community Health Nurs. 2006 Winter;23(4):225-34.
- 12. Kleinman LC, Freeman H, Perlman J, Gelberg L. Homing in on the homeless: assessing the physical health of homeless adults in Los Angeles County using an original method to obtain physical examination data in a survey. Health Serv Res. 1996 Dec;31(5):533-49.
- 13. Lee TC1, Hanlon JG, Ben-David J, Booth GL, Cantor WJ, Connelly PW, Hwang SW. Risk factors for cardiovascular disease in homeless adults. Circulation. 2005 May 24;111(20):2629-35. Epub 2005 May 16.

- 14. Asgary R, Sckell B, Alcabes A, Naderi R, Schoenthaler A, Ogedegbe G. Rates and predictors of uncontrolled hypertension among hypertensive adults using New York City shelter-based clinics. Ann Fam Med. Jan-Feb 2016;14(1):41-6
- 15. Joffres M, Falaschetti E, Gillespie C, Robitallie C, Loustalot F, Poulter N, McAlister FA, Johansen H, Baclic O, Campbell N. Hypertension prevalence, awareness, treatment and control in national surveys from England, the USA and Canada, and correlation with stroke and ischemic heart disease mortality: a cross-sectional study. BMJ Open. 2013 Aug 30;3(8):e003423.doi:10.1136/bmjopen-2013003423.
- 16. Khandor E, Mason K, Chambers C, Rossiter K, Cowan L, Hwang SW. Access to primary health care among homeless adults in Toronto, Canada: results from the Street Health survey. *Open Med* 2011;5(2): e94e103.
- 17. Baggett TP1, Hwang SW, O'Connell JJ, Porneala BC, Stringfellow EJ, Orav EJ, Singer DE, Rigotti NA. Mortality among homeless adults in Boston: shifts in causes of death over a 15-year period. JAMA Intern Med. 2013 Feb 11;173(3):189-95. doi: 10.1001/jamainternmed.2013.1604.
- 18. Hwang SW, Orav EJ, O'Connell JJ, Lebow JM, Brennan TA. Causes of death in homeless adults in Boston. Ann Intern Med. 1997 Apr 15;126(8):625–628.
- 19. Appel LJ, Brands MW, Daniels SR, Karanja N, Elmer PJ, Sacks FM. Dietary approaches to prevent and treat hypertension: a scientific statement from the American Heart Association. *Hypertension*. Feb 2006;47(2):296-308.
- 20. Appel LJ, Champagne CM, Harsha DW, et al. Effects of comprehensive lifestyle modification on blood pressure control: main results of the PREMIER clinical trial. *JAMA*. Apr 23-30 2003;289(16):2083-2093.
- 21. Stamler R, Stamler J, Grimm R, et al. Nutritional therapy for high blood pressure. Final report of a four-year randomized controlled trial--the Hypertension Control Program. *JAMA*. Mar 20 1987;257(11):1484-1491.
- 22. Taylor E, Lake, T., Nysenbaum, J., Peterson, G., Meyers, D. Coordinating Care in the Medical Neighborhood: Critical Components and Available Mechanisms. Agency for Healthcare Research and Quality; 2011. AHRQ Publication No.11-0064. available at <a href="https://pcmh.ahrq.gov/page/coordinating-care-medicalneighborhood-critical-components-and-available-mechanisms">https://pcmh.ahrq.gov/page/coordinating-care-medicalneighborhood-critical-components-and-available-mechanisms</a>
- 23. Pham HH. Good neighbors: how will the patient-centered medical home relate to the rest of the health-care delivery system? *J Gen Intern Med.* Jun;25(6):630-634.
- 24. Gurol-Urganci I, de Jongh T, Vodopivec-Jamsek V, Atun R, Car J. Mobile phone messaging reminders for attendance at healthcare appointments. *Cochrane Database Syst Rev.* 2013, dec 5;2013(12): CD007458. DOI:
- 10.1002/14651858.CD007458.pub3. available at <a href="https://pubmed.ncbi.nlm.nih.gov/24310741/">https://pubmed.ncbi.nlm.nih.gov/24310741/</a>
- 25. Guy R, Hocking J, Wand H, Stott S, Ali H, Kaldor J. How effective are short message service reminders at increasing clinic attendance? A meta-analysis and systematic review. Health Serv Res. 2012 Apr;47(2):614-32.
- 26. Márquez Contreras E1, de la Figuera von Wichmann M, Gil Guillén V, Ylla-Catalá A, Figueras M, Balaña M, Naval J. Effectiveness of an intervention to provide information to patients with hypertension as short text messages and reminders sent to their mobile phone (HTA-Alert)]. Aten Primaria. 2004 Nov 15;34(8):399-405.

- 27. McGillicuddy JW, Gregoski MJ, Weiland AK, Rock RA, Brunner-Jackson BM, Patel SK, Thomas BS, Taber DJ, Chavin KD, Baliga PK, Treiber FA. Mobile Health Medication Adherence and Blood Pressure Control in Renal Transplant Recipients: A Proof-of-Concept Randomized Controlled Trial. JMIR Res Protoc. 2013 Sep 4;2(2):e32.
- 28. Hamine S, Gerth-Guyette E, Faulx D, Green BB, Ginsburg AS. Impact of mHealth chronic disease management on treatment adherence and patient outcomes: a systematic review. J Med Internet Res. 2015 Feb 24:17(2):e52. doi: 10.2196/jmir.3951.
- 29. Dick JJ, Nundy S, Solomon MC, Bishop KN, Chin MH, Peek ME. Feasibility and usability of a text message-based program for diabetes self-management in an urban African-American population. J Diabetes Sci Technol. 2011 Sep 1;5(5):1246-54.
- DeKoekkoek T, Given B, Given CW, Ridenour K, Schueller M, Spoelstra SL.mHealth SMS text messaging interventions and to promote medication adherence: an integrative review. J Clin Nurs. 2015 Oct;24(1920):2722-35. doi: 10.1111/jocn.12918. Epub 2015 Jul 27.
- 31. Marcum ZA, Sevick MA, Handler S. Medication Nonadherence, A diagnosable and Treatable Medical Condition. JAMA, May 2013; 309 (20):2015-6
- 32. Viswanathan M, Golin CE, Jones CD, et al. Interventions to improve adherence to self-administered medications for chronic diseases in the United States: a systematic review. Ann Intern Med. 2012;157(11):785795.
- 33. Post LA, Vaca FE, Doran KM, Luco C, Naftilan M, Dziura J, Brandt C, Bernstein S, Jagminas L, D'Onofrio G. New media use by patients who are homeless: the potential of mHealth to build connectivity. J Med Internet Res. 2013 Sep 3;15(9):e195. doi: 10.2196/jmir.2724.
- 34. Eyrich-Garg KM. Mobile phone technology: a new paradigm for the prevention, treatment, and research of the non-sheltered "street" homeless? J Urban Health. 2010 May;87(3):365-80.
- 35. Asgary R, Sckell B, Alcabes A, Naderi R, Adongo P, Ogedegbe G. Perceptions, attitudes, and experience regarding mHealth among homeless. J Health Commun. 2015;20(12):1473-80
- Jennings L, Lee N, Shore D, Strohminger N, Allison B, Conserve D, Cheskin LJ. US. Minority Homeelss Youth's Access to and Use of Mobile Phones: Implications for Health Intervention Design. J Health Commun. 2016;21(7):725-33
- 37. McInnes DK, Petrakis BA, Gifford AL, Rao SR, Houston TK, Asch STM, O'Toole TP. Retaining Homeless Veterans in Outpatient Care: A Pilot Study of Mobile Phone Text Message Appointment Reminders. AM J Public Health. 2014;104 suppl:s588-94.doi:10.2105/AJPH.2014.302061
- 38. Clover AC, Schueller SM, Winiarski DA, Smith DL, Karnik NS, Zalta A. Automated Mobile Phone-Based Mental Health Resource for Homeelss Youth: Pilot Study Assessing Feasibility and Acceptability. JMIR Ment Health. 2019;6(10):e1511.doi:10.2196/15144
- 39. Foyabo J, Bessetti-Barrett C. Improving clinic attendance through text message reminders to homeless patients with chronic health conditions. 2019, accessed June 2, 2020, available at <a href="https://www.elitecme.com/resource-center/health-information-professionals/improving-clinic-attendancethrough-text-message-reminders-to-homeless-patients-with-chronic-health-conditions/">https://www.elitecme.com/resource-center/health-information-professionals/improving-clinic-attendancethrough-text-message-reminders-to-homeless-patients-with-chronic-health-conditions/</a>
- 40. Prochaska, J. O. & Prochaska, J. M. Helping cure health care systems: Changing minds and behaviour.

Disease Management and Health Outcomes, Medicine, Published 1999, *6*, 335-341, DOI.10.2165/00115677199906060-0004

- 41. Johnson SS, Driskell MM, Johnson JL, Prochaska JM, Zwick W, Prochaska JO. Efficacy of a transtheoretical model-based expert system for antihypertensive adherence. Dis Manag. 2006 Oct;9(5):291301.
- 42. Glasgow RE, Orleans CT, Wagner EH. Does the chronic care model serve also as a template for improving prevention? *Milbank Quarterly.* 2001;79(4):579-612, iv-v.
- 43. Tsai AC, Morton SC, Mangione CM, Keeler EB. A meta-analysis of interventions to improve care for chronic illnesses. *Am J Manag Care*. Aug 2005;11(8):478-488.
- 44. Wagner EH. Chronic disease management: what will it take to improve care for chronic illness? Eff Clin Pract. 1998;1:2-4
- 45. Asgary R, Garland V, Jakubowski A, Sckell B. Colorectal cancer screening among the homeless population of New York City shelter-based clinics. Am J Pub Health. 2014;104(7):1307-13
- 46. Chen ZW, Fang LZ, Chen LY, Dai HL. Comparison of an SMS text messaging and phone reminder to improve attendance at a health promotion center: a randomized controlled trial. J Zhejiang Univ Sci B. 2008 Jan;9(1):34-8.
- 47. Leong KC, Chen WS, Leong KW, Mastura I, Mimi O, Sheikh MA, Zailinawati AH, Ng CJ, Phua KL, Teng CL. The use of text messaging to improve attendance in primary care: a randomized controlled trial. Fam Pract. 2006 Dec;23(6):699-705.
- 48. National Health Care for the Homeless Council. Training and Technical Assistance. Telehealth Webinars, Using Telehealth to manage Diabetes (2020), Tele-Behavioral Health in Homeless Health Care; Why Is it Hard, and What Can we DO About it? (2019), Accessed June 2<sup>nd</sup> 2020, available at <a href="https://nhchc.org/clinical-practice/homeless-services/telehealth/">https://nhchc.org/clinical-practice/homeless-services/telehealth/</a>
- 49. Iheanacho T, Payne K, Tsai J. Mobile, Community-Based buprenorphine Treatment for Veterans Experiencing Homelessness With Opioid Use Disorder: A Pilot, Feasibility Study. Am J Addict. 2020;doi.10.1111/ajad.13055.Online ahead of print
- 50. Gong K, Yan YL, Li Y, Du J, Wang J, Han Y, Zou Y, Z XY, Huang H, She Q. Mobile Health Applications for the Management of Primary Hypertension: A multicenter, Randomized, Controlled Trial. *Medicine*. 2020;99(16):e19715
- 51. How many people experience homelessness? NCH Fact Sheet No. 2. National Coalition for the Homeless Web site. February 2013. (accessed June 2, 2020) http://www.nationalhomeless.org/factsheets/How Many.pdf
- 52. The 2011 Annual Homeless Assessment Report to Congress. Nov 2012. The US Department of Housing and Urban Development Office of Community Planning and Development. (accessed June 2, 2020) <a href="https://www.onecpd.info/resources/documents/2011AHAR">https://www.onecpd.info/resources/documents/2011AHAR</a> FinalReport.pdf
- 53. Project Renewal. What We Do. Accessed June 2, 2020, available at <a href="https://www.projectrenewal.org/programs-overview">https://www.projectrenewal.org/programs-overview</a>
- 54. Whelton PK, Carey RM, Aronow WS et al. 2017

ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice. J Am Coll Cardiol. 2018;71(19):2199-2269. Available at

https://www.onlinejacc.org/content/71/19/2199?\_ga=2.76732177.505114254.15922621811057634203.1592262181

- 55. Bobrow K, Brennan T, Springer D, Levitt NS, Rayner B, Namane M, Yu LM, Tarassenko L, Farmer A. Efficacy of a text messaging (SMS) based intervention for adults with hypertension: protocol for the StAR (SMS Text-message Adherence suppoRt trial) randomised controlled trial. *BMC Public Health*. 2014 Jan 11;14:28. doi: 10.1186/1471-2458-14-28.
- 56. Million Hearts. Tools & Protocols. Accessed June 2, 2020, available at <a href="https://millionhearts.hhs.gov/toolsprotocols/index.html">https://millionhearts.hhs.gov/toolsprotocols/index.html</a>
- 57. Richards AK, Jackson NJ, Cheng EM, Bryg RJ, Brown A, Towfighi A, Sanossian N, Barry F, Li N.

Derivation and Application of a Tool to Estimate Benefits From Multiple Therapies That Reduce Recurrent Stroke Risk. *Stroke*.2020;51(5):1563-1569

- 58. McInnes DK. Self- management Using text Messaging in a Homeless Population. ClinicalTrial.gov. Accessed June 2, 2020, available at https://clinicaltrials.gov/ct2/show/record/NCT03034993
- 59. Guy R, Hocking J, Wand H, Stott S, Ali H, Kaldor J. How effective are short message service reminders at increasing clinic attendance? A meta-analysis and systematic review. Health Serv Res. 2012 Apr;47(2):614-32.

doi: 10.1111/j.1475-6773.2011.01342.x

- 60. Perloff D, Grim C, Flack J, et al. Human blood pressure determination by sphygmomanometry. *Circulation*. Nov 1993;88(5 Pt 1):2460-2470.
- 61. Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. *Med Care*. 1986;24:67–74.
- 62. Morisky D. E., Ang A., Krousel-Wood M, Ward, H. J. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens. 2008;10(5):348-354.
- 63. Lu, M., Safren, S. A., Skolnik, P. R., Rogers, W. H., Coady, W., Hardy, H., & Wilson, I. B. Optimal recall period and response task for self-reported HIV medication adherence. Aids and Behavior, 2008;12(1):86-94. doi:
- 10.1007/s10461-007-9261-4
- 64. Asgary R. Naderi R, Wisnivesky J. Opt-out patient navigation to improve breast and cervical cancer screening among homeless women in New York City shelters and shelter-clinics. J Womens Health (Larchmt). 2017;26(9):999-1003. doi: 10.1089/jwh.2016.6066. [Epub ahead of print].
- 65. Asgary R. Sckell B, Alcabes A, Naderi R, Ogedegbe G. Perspectives of cancer and cancer screening among homeless adults of New York City shelter-based clinics: a qualitative approach. *Cancer Causes Control*, 2015 Oct;26(10):1429-38.
- 66. Collins R, Peto R, MacMahon S, Hebert P, Fiebach NH, Eberlein KA, Godwin J, Qizilbash N, Taylor JO, Hennekens CH. Blood pressure, stroke, and coronary heart disease. Part 2, Short-term reductions in blood

pressure: overview of randomised drug trials in their epidemiological context. Lancet. 1990 Apr 7;335(8693):827-38.

- 67. Lam AY, Fresco P. Medication Adherence Measures: On Overview. Biomed Res Int. 2015; 2015:217074. doi.10.1155/2015/217074
  - 68. Voils CI, King HA, Thorpe CT, et al. Content validity and reliability of a self- report measure of medication nonadherence in hepatitis C treatment. Dig Dis Sci 2019;64:2784–97.
  - 69. Voils CI, King HA, Neelon B, et al. Characterizing weekly self- reported antihypertensive medication nonadherence across repeated occasions. Patient Prefer Adherence 2014;8:643–50.